CLINICAL TRIAL: NCT04272476
Title: The Activation on Prefrontal Cortex With Acupuncture and Moxibustion for Major Depressive Disorder: A Study of Functional Near Infrared Spectroscopy (ACUfNIRS)
Brief Title: The Activation on Prefrontal Cortex With Acupuncture and Moxibustion for Major Depressive Disorder: A Study of Functional Near Infrared Spectroscopy
Acronym: ACUfNIRS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Li ying, Professor, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChengduUTCM
Record Dates: First submitted 2015-03-31; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Depressive Disorder, Major
Keywords: Acupuncture; Moxibustion; Major Depressive Disorder; MDD; Neural Network Reconstruction; cerebral function; functional near infrared spectroscopy (fNIRS) imaging
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acupuncture Therapy; Moxibustion; Fluoxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture and moxibustion (Experimental): Acupuncture points: Baihui(GV 20), Mingmen(GV 4), Bilateral Neiguan(PC 6), Bilateral Shenmen(HT 7), Bilateral Hegu(LI 4), Bilateral Zusanli(ST 36), Bilateral Taichong(LR 3). Each treatment takes about thirty minutes,3 times a week(treatment on Monday, Wednesday and Friday) for 8 weeks.
  Interventions: Other: acupuncture and moxibustion
- Western medicine (Active Comparator): Fluoxetine 20 mg capsule by mouth every day for 8 weeks.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Other: acupuncture and moxibustion
  Arms: Acupuncture and moxibustion
Drug: Fluoxetine
  Other Names: Prozac
  Arms: Western medicine

SUMMARY:
This study evaluates the activation on prefrontal cortex with acupuncture and moxibustion for major depressive disorder.Half of participants will receive the treatment of acupuncture and moxibustion, while the other participants will receive the fluoxetine.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a psychiatric condition with high morbidity, disability, suicide and recurrence rate and become the hot and difficult topics in the medical study. Given the unsatisfactory response rates of many FDA-approved antidepressants, acupuncture is increasingly considered an important alternative therapy. A large number of clinical trials have confirmed that acupuncture is a generally safe, effective, and well-tolerated therapy for depression, but for MDD, the acupuncture clinical trials were only reported out of China. According to the clinical symptoms in patients with MDD, the chief TCM patterns are liver qi constraint and heart yang insufficiency, and the secondary TCM patterns are blood stasis, qi and blood deficiency. So we propose to combine acupuncture with moxibustion and select Baihui (DU20), shenting(DU24), Neiguan (PC6), Hegu (LI4), Taichong (LV3), Zusanli(ST36), Zhongwan (RN 12) and Gaunyuan (RN4) to Soothe the Liver, regulating the heart, warm the yang qi, boost qi and invigorate blood for MDD. We hypothesize that the acupuncture's antidepressant effect is based on the neural network reconstructing mechanism through studying the cerebral cortex function, hippocampal synaptic plasticity, Neurons electrophysiological change. We will employ multi-disciplinary methods in neuropsychology, neuroimaging, computer science, and electrophysiology to explore the important mechanism underlying acupuncture and moxibustion treating MDD.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic criteria of CCMD-3 and DSM-4 depression;
* the score of PHQ-9 should be equal to or more than 15 points; the score of Hamilton Depression Rating Scale should be more than 18 points;
* without any drug treatment over the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The Hamilton score as a measure of depressive degree | 1, 2, 4, 6, 8 weeks after treatment
  Evaluating the patient's depressive degree
The fNIRS score as a measure of prefrontal oxyhemoglobin | 1, 2, 4, 6, 8 weeks after treatment
  Evaluating the patient's prefrontal oxyhemoglobin

OTHER OUTCOMES:
The pHQ-9 score | Screening criteria

CONTACTS AND LOCATIONS:
Overall Officials: Wu Junmei, Doctor, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Teaching Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China